CLINICAL TRIAL: NCT01536730
Title: A Self-Guided Intervention to Promote Condom Use Among African American Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stephanie Sanders, Professor Department of Gender Studies and Associate Director The Kinsey Institute, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R21MH090892-02 (NIH)
Record Dates: First submitted 2011-07-20; First posted 2012-02-22 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Correct Consistent Condom Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homework Intervention Strategy (Experimental)
  Interventions: Behavioral: Homework Intervention Strategy
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Homework Intervention Strategy — Participants assigned to intervention will receive a condom "ditty bag" containing 50 condoms (5 each of 10 types), a variety of 50 lubricants, an instructional DVD, and instructions for the intervention.
  Arms: Homework Intervention Strategy

SUMMARY:
The Centers for Disease Control and Prevention has declared that AIDS is a "state of emergency" in the US for African Americans - young African American men are especially vulnerable in this epidemic. Thus, the development of effective interventions tailored to this population is a national priority. The investigators previous preliminary studies suggest that a brief, clinic-initiated, home-based, self-guided condom use program may effectively promote the acceptance of condom use and increase the quality and consistency of condom-protected sexual behaviors. This pilot study will (1) develop and test the feasibility of this program (Homework Intervention Strategy, HIS) for young African American men attending an urban STD clinic and (2) identify variables that may mediate the efficacy of the program. The HIS has the potential to be readily translated into widespread practice, while requiring only minimal resources. Unlike previously tested interventions, the HIS can be applied to all men who use condoms, regardless of the sex of their partners or their HIV/STI status. To develop the HIS to meet the needs of these high-risk men, the proposed study will include a formative phase during which the basic intervention "instructions" which will be delivered by DVD will be refined and tailored for this population.

One hundred young African American men recruited from an urban STD clinic will be randomized to each of two groups (HIS vs. "standard of care") in a randomized 2-arm trial with 5 assessment periods over the course of 6 months. Assessments will compare the groups on frequency of unprotected sex, quality of the condom use experience, experience of condom use errors and problems, attitudes regarding condom use, condom use acceptability, and condom use self-efficacy and confidence.

ELIGIBILITY:
Inclusion Criteria:

* African American men
* 15 to 24 years of age
* able to read, write and comprehend English
* have engaged penile-vaginal intercourse (PVI) or insertive penile-anal intercourse (PAI) with a partner at least once in the past 30 days
* willing to use a condom
* does not intend to get a partner pregnant in the next 6 months
* consent to participate in the study
* client of the Bell Flower Clinic in Indianapolis, IN in the past 12 months
* has maintained a cell-phone number for the past three months and is willing to use it for data collection and incur fees for voice communication or text messaging it they do not have unlimited plans

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 193 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in number of unprotected sex events at 2 months | 30 days
Change from baseline in number of unprotected sex events at 4 months | 30 days
Change from baseline in number of unprotected sex events at 7 months | 30 days

SECONDARY OUTCOMES:
Change from baseline in condom use errors/problems score as measured by the Condom Use Errors/Problems Survey (CUES) at 2 months. | 30 days
Change from baseline in condom use errors/problems score as measured by the Condom Use Errors/Problems Survey (CUES) at 4 months. | 30 days
Change from baseline in condom use errors/problems score as measured by the Condom Use Errors/Problems Survey (CUES) at 7 months. | 30 days
Change from baseline in self-efficacy for correct condom use score as measured by the Correct Condom Use Self-Efficacy Scale(CCUSES) at 2 months. | 30 days
Change from baseline in self-efficacy for correct condom use score as measured by the Correct Condom Use Self-Efficacy Scale (CCUSES) at 4 months. | 30 days
Change from baseline in self-efficacy for correct condom use score as measured by the Correct Condom Use Self-Efficacy Scale(CCUSES) at 7 months. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie A Sanders, Ph.D., Principal Investigator — Indiana University; William L Yarber, Ph.D., Principal Investigator — Indiana University
Locations (1):
- Bell Flower Clinic, Indianapolis, Indiana, United States